CLINICAL TRIAL: NCT05221411
Title: TAILOR Study: Tacrolimus Versus Mycophenolate for Autolmmune Hepatitis Patients With incompLete Response On First Line Therapy: a Randomized Trial
Brief Title: Tacrolimus Versus Mycophenolate for Autoimmune Hepatitis Patients With Incomplete Response on First Line Therapy
Acronym: TAILOR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Bart van Hoek, Prof. dr., Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P21.089; 2021-003420-33 (EudraCT Number); NL78216.058.21 (Other: CCMO)
Record Dates: First submitted 2022-01-07; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mycofenolate Mofetil (Experimental): Patients in the mycophenolate mofetil (MMF) arm will receive MMF for a total of 12 months (if tolerated)
  Interventions: Drug: Mycophenolate Mofetil
- Tacrolimus (Envarsus) (Experimental): Patients in the tacrolimus (TAC) arm will receive treatment with meltdose TAC for a total of 12 months (if tolerated)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Mycophenolate mofetil will be started at a dose 500mg twice daily. When tolerated and an AUC within range, patients will be titrated to 1000mg twice daily at week two.
  Other Names: Cellcept
  Arms: Mycofenolate Mofetil
Drug: Tacrolimus — Meltdose tacrolimus will be started at a dose of 0.07 mg/kg/day. The drug will be taken orally once-daily in the morning. Dose will be adjusted to reach target AUC and trough levels.
  Other Names: Envarsus
  Arms: Tacrolimus (Envarsus)

SUMMARY:
Rationale: The combination of azathioprine and prednisone is the first-line treatment for autoimmune hepatitis (AIH), a chronic inflammatory disease of the liver. Complete biochemical remission (CR) is the first treatment goal in autoimmune hepatitis. CR is determined by AST and ALT and IgG within the reference range. CR is not reached in a substantial proportion of AIH patients: after one year 50%, after three years around 20% did not achieve CR. Without CR ongoing hepatitis leads to progression towards fibrosis and eventually (decompensated) cirrhosis. Not achieving CR is the most important risk factor for the need for liver transplantation or liver related death, independent of age and presence of cirrhosis. Tacrolimus (TAC) and mycophenolate mofetil (MMF) are frequently used to prevent rejection in kidney and liver transplant patients. In AIH patients with insufficient response or intolerance to first-line therapy in retrospective cohort studies with MMF 0-57% and with TAC 20-95% CR was reached.

Objective: The aim of this study is to compare the effectiveness of TAC with MMF as a second line treatment for AIH. Proportion of patients with CR after 12 months of treatment will be the primary outcome parameter to determine effectivity.

Study design: Randomized open-label two arm study. Patients will be randomized between treatment with TAC or MMF.

Study population: Patients with AIH with an incomplete response (no CR) to first-line treatment are eligible for this study.

Intervention: In the TAC group baseline treatment will be replaced by tacrolimus. In the MMF group baseline treatment will be replaced by MMF. The current dose of prednisolone, or at least 5 mg daily, will be continued in both arms. After achieving CR prednisolone will be tapered according to protocol.

Main study parameters/endpoints: Difference in proportion of patients with CR at 12 months (normalization of ALT, AST and IgG) between the TAC and MMF treatment group.

Secondary parameters:

* Safety and tolerability of TAC and MMF treatments
* Difference in proportion of patients with CR at 6 months (normalization of ALT, AST and IgG) between the TAC and MMF treatment group.
* Difference in ALT, AST and IgG at 6 and 12 months versus baseline
* Difference in fibrogenesis and fibrosis parameters between groups and before and after treatment
* Difference in quality of life between groups and before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Patient is older than 18 years old
* Probable or definite auto immune hepatitis according to the original or simplified IAIHG criteria (>10 points pre-treatment on the original criteria or >6 points on the simplified criteria)(2, 3)
* Incomplete responder on at least a half year of first-line treatment, with at least last 6 months azathioprine / 6-MP) / 6-TG and prednisolone or budesonide, and ALT 1.5 - 10x ULN for at least 2 months
* Patient is capable of understanding the purpose and risks of the study, has been fully informed and has given written informed consent to participate in the study

Exclusion Criteria:

* Presence of decompensated liver disease, defined as ascites, coagulopathy (INR >1.5), encephalopathy, variceal bleed, hepatopulmonal syndrome, hepatorenal syndrome or HCC in the past 6 months
* Signs of other liver diseases as NAFLD, Wilson disease, hemochromatosis, alcoholic liver disease or hepatitis B/C/D
* Clinical diagnosis of overlap / variant syndrome with PBC or PSC
* Liver transplantation in the medical history or currently on the waiting list for liver transplantation
* Incompliance with therapy during the last 12 months
* Active infections during inclusion including latent tuberculosis and HIV co-infection
* Allergic or hypersensitive to tacrolimus or MMF
* An estimated glomerular filtration rate (eGFR) of <60 mL/min
* Pregnancy or intention to become pregnant in the next 12 months
* Use of TAC or MMF in the past
* Malignancy in the medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Complete biochemical remission | 52 weeks
  The proportion of patients with CR after 12 months of treatment with TAC compared to MMF in patients with AIH with an incomplete response to first-line treatment.

SECONDARY OUTCOMES:
Safety and Tolerability | 52 weeks
  Number and severity of side effects; Rate of stopping treatment due to side effects; serum creatinin & potassium; Blood pressure; Blood glucose levels and incidence of new onset diabetes; Number of (opportunistic) infections; tremor; diarrhea
Proportion of patients with complete biochemical remission after 6 months | 24 weeks
  Defined as ALT, AST and IgG below the upper limit of normal
Proportion of patients with partial response | 52 weeks
  defined as decrease of AST and ALT, but no normalization
Proportion of patients with insufficient treatment response | 52 weeks
  less than 25% reduction in ALT after 6 and 12 months treatment
Dose reduction of prednisone | 52 weeks
  Difference between dose at inclusion and dose at the end of study
Cessation rate of prednisone | 52 weeks
  The number of patients able to completely withdraw from corticosteroids
Change of AST | 24 and 52 weeks
  at 6 and 12 months versus baseline and between groups at the same time points
Change of ALT | 24 and 52 weeks
  at 6 and 12 months versus baseline and between groups at the same time points
Change of IgG | 24 and 52 weeks
  at 6 and 12 months versus baseline and between groups at the same time points
Liver function | 24 and 52 weeks
  Total bilirubin, albumin, INR and MELD-score after 6 and 12 months between groups
Fibrosis | 52 weeks
  Liver stiffness as measured by elastography and blood fibrosis markers (ELF)
Influence of liver disease on the quality of life | 52 weeks
  using the validated liver disease symptom index (LDSI)
Treatment effect on health status | 52 weeks
  using the validated EQ5D
Cost-effectiveness based on empiric data obtained by this study. | 52 weeks
  Economic evaluation including a cost-effectiveness evaluation
Cost-effectiveness from a societal perspective | 52 weeks
  Economic evaluation including a cost-utility evaluation (costs per QALY)

CONTACTS AND LOCATIONS:
Overall Officials: Bart van Hoek, Principal Investigator — Leiden University Medical Center
Locations (6):
- Netherlands (6):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Reinier de Graaf Gasthuis, Delft
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center +, Maastricht
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stoelinga AEC, Tushuizen ME, van den Hout WB, Girondo MDMR, de Vries ES, Levens AD, Moes DAR, Gevers TJG, van der Meer S, Brouwer HT, de Jonge HJM, de Boer YS, Beuers UHW, van der Meer AJ, van den Berg AP, Guichelaar MMJ, Drenth JPH, van Hoek B; Dutch Autoimmune Hepatitis Group. Tacrolimus versus mycophenolate for AutoImmune hepatitis patients with incompLete response On first-line therapy (TAILOR study): a study protocol for a phase III, open-label, multicentre, randomised controlled trial. Trials. 2024 Jan 17;25(1):61. doi: 10.1186/s13063-023-07832-w. PMID 38233878